CLINICAL TRIAL: NCT02001441
Title: Physical Activity Levels and Hippocampal Sub-region Structure in MCI
Brief Title: UCLA Fitness and Memory Study of Activity In Mild Cognitive Impairment (AIM)
Acronym: AIM
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David Merrill, MD, PhD, Assistant Professor, University of California, Los Angeles
Other Study IDs: 13-000781; UL1TR000124 (NIH)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Physical Activity, Aging, Memory, Cognitive Impairment, MRI, Neuroscience
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
This project will examine the relationship between physical activity levels, brain structure and memory function in adults with Mild Cognitive Impairment (MCI) aged 60 to 75. The study will follow 30 adults with age-associated memory impairment or MCI over the course of 18 months. During this time, subjects' physical activity levels will be measured regularly and related to both the thickness their hippocampus and to their memory performance. Subjects will be recruited and screened for major health problems at UCLA. Physical activity will be tracked for two weeks using accelerometers at baseline and every 6 months during the study. At baseline and at the end of the study, subjects will undergo a structural MRI brain scan to measure hippocampal thickness, as well as a neuropsychological evaluation to measure memory function. The study will seek to determine the relationship between physical activity level, hippocampal thickness and memory performance in older adults with age-associated memory impairment.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the study
* 60-89 years of age
* Diagnostic criteria for Mild Cognitive Impairment diagnosis: subjective memory complaints, Montreal Cognitive Assessment score of <26, intact instrumental activities of daily living (Smith et al., 1996) OR subjective age-associated memory complaints
* Cohabitation with an adult capable of ensuring correct usage of the physical activity monitors during the study and verifying self-reports of activity levels.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Screening laboratory tests and EKG without significant abnormalities that might interfere with the study. If screening laboratory tests or EKG show abnormalities, PI may request clearance from primary care physician before subject continues in study.

Exclusion Criteria:

* Comorbid conditions impacting mobility
* Current, untreated depression: BDI-II score >13
* Diagnosis of probable Alzheimer's disease (AD) or any other dementia (e.g., vascular, Lewy body, frontotemporal).
* Evidence of other neurological or physical illness that can produce cognitive deterioration. Volunteers with a history of head trauma, stroke, TIA, carotid bruits, or lacunes on MRI scans will be excluded.
* Contraindication to the MRI including claustrophobia, metal in body, surgery within 60 days, certain medical implants or previous abnormal MRI results.
* History of cardiovascular disease
* Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100)
* Current diagnosis of any major psychiatric disorder according to the DSM-IV TR criteria (APA, 2000), including current alcoholism or substance addiction.
* Current use of marijuana
* Previous use of marijuana for at least 15 days in a month, initiating use during adolescence and continuing for at least one year

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Southern California Residents with memory complaints aged 60-89.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Activity level correlation with hippocampal thickness | 18 months
  Correlation of activity levels, as measured using ankle accelerometers, with hippocampal thickness, as measured using brain Magnetic Resonance Imaging (MRI).

SECONDARY OUTCOMES:
Activity level correlation with memory performance | 18 months
  Correlation of activity levels, as measured using ankle accelerometers, with memory performance, as measured by neuropsychological evaluations

OTHER OUTCOMES:
Baseline measures prediction of follow-up measures | 18 months
  Change in ankle accelerometer, brain MRI and neuropsychological data from baseline to 18 months
Activity level correlation with other measures controlling for other factors | 18 months
  Changes in ankle accelerometer data compared to changes in brain MRI and neuropsychological data from baseline to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David Merrill, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Longevity Center, Los Angeles, California, United States

REFERENCES:
- See also: Longevity Center Research Laboratory — http://www.semel.ucla.edu/longevity/research